CLINICAL TRIAL: NCT06333223
Title: Polyphenols and Probiotics to Improve Menopausal Symptoms Via the Gut-Brain Axis
Acronym: SYMPTOGUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Collaborators: King's College (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Prof, University of Roehampton
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: LSC 23/ 396
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-03

CONDITIONS: Menopause
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Arm 1: Mixture of (Poly)phenols and a probiotic supplement Arm 2: (Poly)phenols and maltodextrin (placebo)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixture of (Poly)phenols and a probiotic supplement (Experimental): This is a Mixture of (Poly)phenols and a probiotic supplement
  Interventions: Dietary Supplement: Mixture of (Poly)phenols and a probiotic supplement
- (Poly)phenols and maltodextrin (Placebo Comparator): This is a mixture of (Poly)phenols and maltodextrin (placebo comparator)
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Mixture of (Poly)phenols and a probiotic supplement — Mixture of (Poly)phenols and a probiotic supplement
  Arms: Mixture of (Poly)phenols and a probiotic supplement
Dietary Supplement: Placebo comparator — Mixture of (Poly)phenols and a placebo maltodextrin comparator
  Other Names: (Poly)phenols and maltodextrin
  Arms: (Poly)phenols and maltodextrin

SUMMARY:
Menopause is one of the most significant lifecourse challenges for women. The decline in female sex hormones, in particular estrogen, during menopause leads to an increased risk in cardiometabolic diseases, and a decrease in quality of life due to symptoms such as low mood, anxiety, hot flushes and difficulty sleeping. As life expectancy continues to increase, on average, women will spend one third of their life in the postmenopausal period. Increasing evidence suggests that the gut microbiota plays a key role in menopause-related symptoms and conditions, being one of the main regulators of circulating sex hormones. Menopause has been linked to gut dysbiosis and lower gut microbial diversity, therefore nutritional strategies targeting the gut microbiome may be an effective approach to improve women's health during menopause. Both (poly)phenols and probiotics are promising candidates for the prevention and treatment of menopausal symptoms via different mechanisms, including the modulation of the gut-brain axis, while emerging evidence indicates that using both together may be a better approach than traditional carbohydrate-based synbiotics.

To our knowledge, the efficacy of a (poly)phenol based synbiotic targeting the gut microbiome for improvement of menopausal symptoms has not been investigated so far.

DETAILED DESCRIPTION:
The main aim of this work is to investigate whether a combination of (poly)phenols and probiotics will improve mood, anxiety and other menopausal symptoms via a gut microbiota related mechanism. This is a double-blind randomized crossover study with a total of 30 postmenopausal women (i.e participants will be divided into two groups with 15 participants in each group) and will test the effects of 8-week daily consumption of either a combination of a (poly)phenol supplement specifically designed to target the gut microbiota and a probiotic supplement specifically designed to target the gut-brain axis or the the (poly)phenol supplement and maltodextrin (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Adults >48 years
* Post-menopausal female subjects without clinical signs or symptoms of cardiovascular disease, no menstruation cycle for more than 1 year, postmenopausal status conformed by female hormone analysis
* For intervention purposes, eligible participants are also required to have a mobile phone and be able to read and speak English.

Exclusion Criteria:

* • People with comorbid conditions that may limit participation in the study, such as a history of an acute cardiovascular event, uncontrolled hypertension, cancer or major psychiatric or cognitive problems

  * People who are already participating in a weight loss programme
  * People receiving drug treatment for lipid metabolisms (e.g., statins
  * People with a history of long-term use of medicines known to influence glucose metabolism (e.g., corticosteroids)
  * People who take antibiotics or bacterial agents (Probiotics) within 1 month
  * Pregnant women, women ready for pregnancy, and nursing mothers
  * Post-menopausal female subjects without clinical signs or symptoms of cardiovascular disease
  * acute inflammation
  * cardiac arrhythmia
  * renal failure
  * heart failure (NYHA II-IV)
  * diabetes mellitus
  * C-reactive protein > 0.5 mg/dL
  * malignant disease
  * hypotension (≤100 / 60 mm Hg)
  * Women who require hormone replacement therapy during the development of the protocol.

Ages: 48 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menopause Female Women
Enrollment: 30 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in blood chemistry levels | Change from baseline to 8 and 16 weeks of the intervention
  To investigate whether a combination of (poly)phenols and probiotics intervention lowers the blood chemitry parameters compared to the baseline

SECONDARY OUTCOMES:
Change in BMI (body mass index) Scores | Change from baseline to 8 and 16 weeks of the intervention
  To test whether a combination of (poly)phenols and probiotics intervention affect body mass index express in kg/m^2
Change in the gut microbiota diversity | Change from baseline to 8 and 16 weeks of the intervention
  To test whether a combination of (poly)phenols and probiotics intervention impact on the faecal microbiota composition and microbial composition express as ratio compared to the baseline levels
Change in dietary habits | Change from baseline to 8 and 16 weeks of the intervention
  To test whether a combination of (poly)phenols and probiotics intervention impact an assessment of dietary intake in the study population using a validated four-day food diary compared to the baseline levels
Change in Quality IPAQ | Change from baseline to 8 and 16 weeks of the intervention
  To test whether a combination of (poly)phenols and probiotics intervention impact an assessment of physical activity questionnaire in the study population using a validated four-day food diary compared to the baseline levels
Change in inflammatory biomarkes | Change from baseline to 8 and 16 weeks of the intervention
  To test whether a combination of (poly)phenols and probiotics intervention impact CRP, IL10,IL-6 and INFY levels in the study population using ELISA immunoassays compared to the baseline levels

CONTACTS AND LOCATIONS:
Overall Officials: ADELE COSTABILE, Study Director — University of Roehampton
Locations (2):
- United Kingdom (2):
  - Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK
  - Adele Costabile, London

IPD SHARING:
Plan to Share IPD: No